CLINICAL TRIAL: NCT03138473
Title: Impact of Residual Syntax Score and Syntax Revascularization Index on Outcomes of Acute Coronary Syndrome Patients With Multi-Vessel Disease
Brief Title: Impact of Residual Syntax Score and Syntax Revascularization Index on Outcomes of ACS Patients With Multi-Vessel Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Abdelbadee Abdelhameed Othman, Resident Physician, Assiut University
Other Study IDs: 17100078
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Multi Vessel Coronary Artery Disease; NSTEMI - Non-ST Segment Elevation MI; ACS - Acute Coronary Syndrome
Keywords: SYNTAX Score; residual SYNTAX score; SYNTAX Revascularization Index
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Group: Acute Coronary Syndrome Patients With Multi-Vessel Disease. The Residual SYNTAX score (rSS) and the SYNTAX Revascularization Index (SRI) will be calculated in this group and its relationship with patient outcomes either in hospital or in 6 months to 1 year follow-up will be evaluated.
  Interventions: Diagnostic Test: Residual SYNTAX Score; Diagnostic Test: SYNTAX Revascularization Index

INTERVENTIONS:
Diagnostic Test: Residual SYNTAX Score — The baseline SYNTAX score and the residual SYNTAX score (rSS) are calculated by summing up the individual scores for each lesion with a diameter stenosis ≥50% in vessels with a diameter ≥ 1.5 mm in the angiography obtained before and after the procedure. The SYNTAX algorithm of scoring is fully described elsewhere.
  The modified Age, Creatinine, and Ejection Fraction (ACEF) score is calculated based on the age, creatinine clearance (CrCl) and left ventricular ejection fraction (LVEF), using the formula age/LVEF +1 point for every 10 ml/min/1.73 m2 reduction of CrCl below 60 ml/min/1.73 m2 (1 point for CrCl between 59 and 50, 2 points for CrCl between 49 and 40 and 3 points for CrCl between 39 and 30 ml/min/1.73 m2). The CrCl is calculated via the Cockroft-Gault equation using age, gender weight and serum creatinine before PCI. The baseline SYNTAX score was then multiplied by the modified ACEF score to obtain the baseline clinical SYNTAX score.
Diagnostic Test: SYNTAX Revascularization Index — The SYNTAX Revascularization Index (SRI), representing the proportion of CAD burden treated by PCI, was calculated using the following formula: SRI= (1-[rSS/bSS]) ×100.

SUMMARY:
The investigators want to assess the use of the residual SYNTAX score and the SYNTAX Revascularization Index as predictors for in-hospital outcomes and mid-term (6 months to 1 year) outcomes in patients with multi-vessel disease (MVD) who undergo PCI in the setting of STEMI or NSTEACS. Both values will be calculated in a number of patients over one year, and the relationship between both values and patient outcomes will be evaluated.

DETAILED DESCRIPTION:
Significant non-culprit coronary stenosis is noted in 40-70% of patients with ST-elevation Myocardial Infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI). Presence of multivessel disease (MVD) has been associated with poorer clinical outcomes. MVD in STEMI may confer an increased risk of recurrent ischemia and mortality. However, the impact of MVD on prognosis in STEMI may vary depending on the characteristics of coronary artery disease (CAD) present.

Current guidelines recommend that only the infarct-related artery should be treated. However, RCTs have suggested that a strategy of multivessel PCI, either at the time of primary PCI or as a planned, staged procedure, may be beneficial and safe in selected patients with STEMI. On the basis of these findings, the prior Class III (Harm) recommendation with regard to multivessel primary PCI in hemodynamically stable patients with STEMI has been upgraded and modified to a Class IIb recommendation to include consideration of multivessel PCI, either at the time of primary PCI or as a planned, staged procedure.

Early invasive treatment in high-risk patients with non-ST-elevation acute coronary syndrome (NSTEACS) has been shown to improve their prognosis in terms of cardiovascular death and reinfarction. The prevalence of multivessel disease in these patients stands at about 50% and experts agree that performing complete revascularization is beneficial in such patients.

Accordingly, the SYNergy between PCI with TAXus and cardiac surgery (SYNTAX) score has been developed in 2005 in Erasmus Medical Center in the Netherlands to evaluate the severity of coronary artery disease in the settings of left main or MVD.

The investigators have observed a growing interest in residual disease burden after PCI. The residual SYNTAX score (rSS), described by Genereux and colleagues is a strong prognostic factor of coronary events and all-cause death in patients who have undergone PCI. This score has subsequently been validated by other groups and been shown to have good prognostic accuracy for adverse ischemic outcomes after PCI.

The SYNTAX Revascularisation Index (SRI), which takes into account the severity and extent of baseline CAD (as assessed by the baseline SYNTAX score [bSS]) and the residual CAD after PCI (as assessed by the rSS) has been used in determining the proportion of CAD that has been treated, and has been shown to have prognostic utility in PCI for MVD.

Here, the investigators want to assess the use of the residual SYNTAX score and the SYNTAX Revascularization Index as predictors for in-hospital outcomes and mid-term (up to two year) outcomes in patients with multi-vessel disease (MVD) who undergo PCI in the setting of STEMI or NSTEACS.

ELIGIBILITY:
Inclusion Criteria:

* All ACS (STEMI and NSTEACS) patients undergoing PCI in the setting of MVD.

Exclusion Criteria:

* Patients receiving fibrinolytic therapy.
* Patients with cardiogenic shock
* Post-CABG patients
* Patients with severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to the Assiut University Hospitals Department of Cardiology will be collected over one year starting 1st of July 2017 till 30th of June 2018.
  Considering the primary end-point of the study (MACE rate 28%) (Khan et al, 2016), the estimated sample size of the population, based on power of 85%, and alpha= 5%, is calculated to be = 108 patients.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
In-hospital major adverse cardiac events (MACE) | 2 Years
  A composite of cardiac death (including periprocedural), non-fatal myocardial infarction, congestive heart failure, unplanned revascularization including target vessel revascularization (TVR), target lesion revascularization (TLR) and Coronary artery bypass graft (CABG).

SECONDARY OUTCOMES:
The individual components of the primary end-point | 2 Years
  Cardiac death (including periprocedural), non-fatal myocardial infarction, congestive heart failure, unplanned revascularization including target vessel revascularization (TVR), target lesion revascularization (TLR) and Coronary artery bypass graft (CABG)
Major Bleeding | 2 Years
  ACUITY defined major bleeding (Stone et al, 2004)
Acute kidney injury (AKI) | 2 Years
  a 25% relative or 0.5mg/dL (44.2µmol/L) absolute increase in presenting serum creatinine after PPCI.
6 months- 1 year MACE, and its individual components. | 2 Years
  Cardiac death (including periprocedural), non-fatal myocardial infarction, congestive heart failure, unplanned revascularization including target vessel revascularization (TVR), target lesion revascularization (TLR) and Coronary artery bypass graft (CABG),and a composite of these components.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa R. Dimitry, MD, Study Chair — Department of Cardiology, Assiut University Faculty of Medicine; Tarek A. Nagib, MD, Study Director — Department of Cardiology, Assiut University Faculty of Medicine; Khaled M. Elmaghraby, MD, Study Director — Department of Cardiology, Assiut University Faculty of Medicine
Locations (1):
- Assiut University Heart Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Boden H, Velders MA, van der Hoeven BL, Cannegieter SC, Schalij MJ. In-hospital major bleeding and its clinical relevance in patients with ST elevation myocardial infarction treated with primary percutaneous coronary intervention. Am J Cardiol. 2013 Nov 15;112(10):1533-9. doi: 10.1016/j.amjcard.2013.06.025. Epub 2013 Aug 14. PMID 23953696
- [Background] Claessen BE, Dangas GD, Weisz G, Witzenbichler B, Guagliumi G, Mockel M, Brener SJ, Xu K, Henriques JP, Mehran R, Stone GW. Prognostic impact of a chronic total occlusion in a non-infarct-related artery in patients with ST-segment elevation myocardial infarction: 3-year results from the HORIZONS-AMI trial. Eur Heart J. 2012 Mar;33(6):768-75. doi: 10.1093/eurheartj/ehr471. Epub 2012 Jan 12. PMID 22240495
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Background] Farooq V, Serruys PW, Bourantas CV, Zhang Y, Muramatsu T, Feldman T, Holmes DR, Mack M, Morice MC, Stahle E, Colombo A, de Vries T, Morel MA, Dawkins KD, Kappetein AP, Mohr FW. Quantification of incomplete revascularization and its association with five-year mortality in the synergy between percutaneous coronary intervention with taxus and cardiac surgery (SYNTAX) trial validation of the residual SYNTAX score. Circulation. 2013 Jul 9;128(2):141-51. doi: 10.1161/CIRCULATIONAHA.113.001803. Epub 2013 Jun 13. PMID 23766350
- [Background] Fox KA, Clayton TC, Damman P, Pocock SJ, de Winter RJ, Tijssen JG, Lagerqvist B, Wallentin L; FIR Collaboration. Long-term outcome of a routine versus selective invasive strategy in patients with non-ST-segment elevation acute coronary syndrome a meta-analysis of individual patient data. J Am Coll Cardiol. 2010 Jun 1;55(22):2435-45. doi: 10.1016/j.jacc.2010.03.007. Epub 2010 Mar 30. PMID 20359842
- [Background] Garg S, Sarno G, Garcia-Garcia HM, Girasis C, Wykrzykowska J, Dawkins KD, Serruys PW; ARTS-II Investigators. A new tool for the risk stratification of patients with complex coronary artery disease: the Clinical SYNTAX Score. Circ Cardiovasc Interv. 2010 Aug;3(4):317-26. doi: 10.1161/CIRCINTERVENTIONS.109.914051. Epub 2010 Jul 20. PMID 20647561
- [Background] Genereux P, Campos CM, Yadav M, Palmerini T, Caixeta A, Xu K, Francese DP, Dangas GD, Mehran R, Leon MB, Serruys PW, Stone GW. Reasonable incomplete revascularisation after percutaneous coronary intervention: the SYNTAX Revascularisation Index. EuroIntervention. 2015 Oct;11(6):634-42. doi: 10.4244/EIJY14M10_05. PMID 25308300
- [Background] Genereux P, Palmerini T, Caixeta A, Rosner G, Green P, Dressler O, Xu K, Parise H, Mehran R, Serruys PW, Stone GW. Quantification and impact of untreated coronary artery disease after percutaneous coronary intervention: the residual SYNTAX (Synergy Between PCI with Taxus and Cardiac Surgery) score. J Am Coll Cardiol. 2012 Jun 12;59(24):2165-74. doi: 10.1016/j.jacc.2012.03.010. Epub 2012 Apr 4. PMID 22483327
- [Background] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Background] Hoebers LP, Vis MM, Claessen BE, van der Schaaf RJ, Kikkert WJ, Baan J Jr, de Winter RJ, Piek JJ, Tijssen JG, Dangas GD, Henriques JP. The impact of multivessel disease with and without a co-existing chronic total occlusion on short- and long-term mortality in ST-elevation myocardial infarction patients with and without cardiogenic shock. Eur J Heart Fail. 2013 Apr;15(4):425-32. doi: 10.1093/eurjhf/hfs182. Epub 2012 Nov 12. PMID 23148116
- [Background] Khan R, Al-Hawwas M, Hatem R, Azzalini L, Fortier A, Joliecoeur EM, Tanguay JF, Lavoie-L'Allier P, Ly HQ. Prognostic impact of the residual SYNTAX score on in-hospital outcomes in patients undergoing primary percutaneous coronary intervention. Catheter Cardiovasc Interv. 2016 Nov;88(5):740-747. doi: 10.1002/ccd.26413. Epub 2016 Feb 1. PMID 26833916
- [Background] Lee JH, Park HS, Chae SC, Cho Y, Yang DH, Jeong MH, Kim YJ, Kim KS, Hur SH, Seong IW, Hong TJ, Cho MC, Kim CJ, Jun JE, Park WH; Korea Acute Myocardial Infarction Registry Investigators. Predictors of six-month major adverse cardiac events in 30-day survivors after acute myocardial infarction (from the Korea Acute Myocardial Infarction Registry). Am J Cardiol. 2009 Jul 15;104(2):182-9. doi: 10.1016/j.amjcard.2009.03.010. PMID 19576343
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Stone GW, Bertrand M, Colombo A, Dangas G, Farkouh ME, Feit F, Lansky AJ, Lincoff AM, Mehran R, Moses JW, Ohman M, White HD. Acute Catheterization and Urgent Intervention Triage strategY (ACUITY) trial: study design and rationale. Am Heart J. 2004 Nov;148(5):764-75. doi: 10.1016/j.ahj.2004.04.036. PMID 15523305
- [Background] Toma M, Buller CE, Westerhout CM, Fu Y, O'Neill WW, Holmes DR Jr, Hamm CW, Granger CB, Armstrong PW; APEX-AMI Investigators. Non-culprit coronary artery percutaneous coronary intervention during acute ST-segment elevation myocardial infarction: insights from the APEX-AMI trial. Eur Heart J. 2010 Jul;31(14):1701-7. doi: 10.1093/eurheartj/ehq129. Epub 2010 Jun 8. PMID 20530505
- [Background] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Background] Wykrzykowska JJ, Garg S, Onuma Y, de Vries T, Goedhart D, Morel MA, van Es GA, Buszman P, Linke A, Ischinger T, Klauss V, Corti R, Eberli F, Wijns W, Morice MC, di Mario C, van Geuns RJ, Juni P, Windecker S, Serruys PW. Value of age, creatinine, and ejection fraction (ACEF score) in assessing risk in patients undergoing percutaneous coronary interventions in the 'All-Comers' LEADERS trial. Circ Cardiovasc Interv. 2011 Feb 1;4(1):47-56. doi: 10.1161/CIRCINTERVENTIONS.110.958389. Epub 2011 Jan 4. PMID 21205944